CLINICAL TRIAL: NCT01343394
Title: Safety of Autologous Human Umbilical Cord Blood Mononuclear Fraction to Treat Acquired Hearing Loss in Children
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: UT-IRB insists on protocol design change -Not rel to any pt. safety/non-compliance-Recruiting halted at UT/MHHS but may resume at FLHosp for Children-OrlandoFL
Sponsor: Aryn Knight (Other)
Collaborators: Cord Blood Registry, Inc. (Industry); The University of Texas Health Science Center, Houston (Other); M.D. Anderson Cancer Center (Other); Baylor College of Medicine (Other); The Methodist Hospital Research Institute (Other); Florida Hospital for Children (Other)
Responsible Party: Sponsor-Investigator, Aryn Knight, AVP Research, Memorial Hermann Health System
Organization: Memorial Hermann Health System (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JB IND14312
Record Dates: First submitted 2011-04-25; First posted 2011-04-28 (Estimated); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Hearing Loss
Keywords: Autologous; Stem Cells; Hearing Loss; Children
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Biologic; Autologous Cell Injection (Experimental)
  Interventions: Biological: Autologous Human Umbilical Cord Blood

INTERVENTIONS:
Biological: Autologous Human Umbilical Cord Blood — 6 million cells/kg will be administered intravenously at one treatment time point.
  Other Names: Autologous Human Umbilical Cord Blood Mononuclear Fraction Cells; Patient's Own Stem Cells

SUMMARY:
The objectives of this study are:

1. To see if autologous human umbilical cord blood treatment is safe for children with acquired hearing loss, and
2. To determine if late functional outcome is improved following autologous human umbilical cord blood treatment for children with acquired hearing loss.

DETAILED DESCRIPTION:
Acquired sensorineural hearing loss is characterized by a loss of functioning hair cells in the Organ of Corti, with greater hair cell loss correlating with more severe hearing impairment. Children with sensorineural hearing loss experience difficulty developing normal language which usually leads to poor academic and social development. Currently, there are no reparative therapeutic options available, and treatments are designed to augment the diminished function of the injured Organ of Corti.

Pre-clinical data suggest progenitor cell infusions may enhance intrinsic repair mechanisms in the Organ of Corti which may restore hair cells. This treatment could ultimately lead to hearing improvement. Human umbilical cord blood (hUCB) is an available, autologous, stored progenitor cell population available for potential therapeutic use. The primary objective of this study is to determine the safety of autologous hUCB infusion in children with acquired hearing loss. The secondary objective is to determine if functional, physiologic and anatomic outcomes are improved following hUCB treatment in this patient population.

ELIGIBILITY:
Inclusion Criteria:

1. Evidence of a moderate to profound sensorineural hearing loss.
2. Normally shaped cochlea, as determined by MRI.
3. The loss must be considered acquired, NOT syndromic.
4. The patient must be fitted for hearing aids of the detection of the loss.
5. Enrollment in a parent/child intervention program.
6. Between 6 weeks and 18 months of age at the time of cord blood infusion.
7. Ability of child and caregiver to travel to Houston for treatment and all follow-up appointments. (Patient's family is responsible for the cost of travel to and lodging in Houston).

Exclusion Criteria:

1. Inability to obtain pertinent medical records.
2. Known history or

   * Recently treated ear or other infection.
   * Renal disease.
   * Hepatic disease.
   * Malignancy.
   * HIV.
   * Immunosuppression (WBC < 3,000).
   * Evidence of an extensive stroke (> 100ml).
   * Pneumonia, or chronic lung disease.
3. hUCB sample contamination.
4. Participation in a concurrent intervention study.
5. Desire for organ donation in the event of death.
6. Unwillingness or inability to stay 4 days following hUCB infusion, and to return for the one month, six month and one year follow-up visits.
7. Presence of a cochlear implant device.
8. Evidence of a syndrome.
9. Positive test for genetic hearing loss.
10. Evidence of conductive hearing loss.
11. Documented evidence of recurrent middle ear infections (> 5/year).
12. Otitis media at the time of examination.
13. Mild sensorineural hearing loss.
14. Over 18 months at the time of infusion.

Ages: 6 Weeks to 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2011-04; Primary Completion 2013-01 (Actual); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
Physiologic Outcome | One year
  Age appropriate physiologic outcome measures will be recorded pre-treatment, and one year following hUCB treatment

SECONDARY OUTCOMES:
Functional Outcome | one year
  Age appropriate Speech-Language assessments will be performed pre-treatment and one year post-treatment.

CONTACTS AND LOCATIONS:
Overall Officials: James E. Baumgartner, MD, Principal Investigator — MHHS, Houston,TX & FL Hospital for Children, Orlando, FL; Linda S. Baumgartner, CCC-SLP, LSLS CERT.AVT, Principal Investigator — Speech Therapists for Children; Samir Fakhri, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- Children's Memorial Hermann Hospital, Houston, Texas, United States